CLINICAL TRIAL: NCT00797966
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study of the Safety and Efficacy of OPC-34712 as Adjunctive Therapy in the Treatment of Patients With Major Depressive Disorder
Brief Title: Study of the Safety and Efficacy of OPC-34712 as Adjunctive Therapy in the Treatment of Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 331-08-211
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Major Depressive Disorder
Keywords: OPC-34712, Major Depressive Disorder, Adjunctive Treatment
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram; Fluoxetine; Paroxetine; Sertraline; Desvenlafaxine Succinate; Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): OPC-34712 + ADT
  Interventions: Drug: OPC-34712; Drug: ADT
- 2 (Placebo Comparator): Placebo + ADT
  Interventions: Drug: Placebo; Drug: ADT

INTERVENTIONS:
Drug: OPC-34712 — Tablets, Oral, 1 - 4 mg OPC-34712 variable dose once daily, 14 weeks
  Other Names: Generic Name: Brexpiprazole
  Arms: 1
Drug: Placebo — Tablets, Oral, 1- 4 mg OPC-34712 once daily, 14 weeks
  Arms: 2
Drug: ADT — Tablets, 10 - 225 mgs, dose once daily, 14 weeks
  Other Names: Each individual will receive one of the following 6 ADTs:; Escitalopram (Lexapro); Fluoxetine (Prozac); Paroxetine CR (Paxil CR); Sertraline (Zoloft); Desvenlafaxine (Pristiq); Venalfaxine XR (Effexor XR)

SUMMARY:
Primary: To compare the efficacy of OPC-34712 to placebo as adjunctive treatment to an assigned open-label marketed antidepressant treatment (ADT)in patients who demonstrate an incomplete response to a prospective eight week trial of the same assigned open-label marketed ADT.

DETAILED DESCRIPTION:
A comparison of the Fixed dose arm (OPC-31712, 0.15 mg) verses placebo was included as a general secondary efficacy variable and results for this dose group comparison are included under each of the Outcome Measures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 65 years of age, with diagnosis of major depressive disorder, as defined by DSM-IV-TR criteria
* The current depressive episode must be equal to or greater than 8 weeks in duration
* Subjects must report a history for the current depressive episode of an inadequate response to at least one and no more than three adequate antidepressant treatments.

Exclusion Criteria:

* Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving study drug.
* Subjects who report an inadequate response to more than three adequate trials of antidepressant treatments during current depressive episode at a therapeutic dose for an adequate duration.
* Subjects with a current Axis I (DSM-IV-TR) diagnosis of:

  * Delirium, dementia,amnestic or other cognitive disorder
  * Schizophrenia, schizoaffective disorder, or other psychotic disorder
  * Bipolar I or II disorder
  * Subjects with a clinically significant current Axis II (DSM-IV-TR)
  * diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal or histrionic personality disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (50):
- United States (50):
  - Pacific Clinical Research Medical Group, Arcadia, California
  - Southwestern Research, Beverly Hills, California
  - Synergy Escondido, Escondido, California
  - Collaborative Neuroscience Network Inc., Garden Grove, California
  - Synergy Clinical Research Center, National City, California
  - Excell Research, Oceanside, California
  - Affiliated Research Institute, San Diego, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - Radiant Research Center, Denver, Colorado
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - CNS Clinical Research Group, Coral Springs, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Accurate Clinical Trials, Kissimee, Florida
  - Clinical Neurosciences Solutions, Orlando, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - University of South Florida College of Medicine Psychiatry Center, Tampa, Florida
  - Janus Center, West Palm Beach, Florida
  - Carman Research, Smyrna, Georgia
  - Uptown Research Institute, Chicago, Illinois
  - Midwest Center for Neurobehavioral Medicine, Oakbrook Terrace, Illinois
  - The Davis Clinic, PC, Indianapolis, Indiana
  - Vince & Associates Clinical Research, Overland Park, Kansas
  - Pharmasite Research, Inc., Baltimore, Maryland
  - Bioscience Research, Mount Kisco, New York
  - Eastside Comprehensive Medical Center, New York, New York
  - Medical & Behavioral Health Research, PC, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Carolinas HealthCare - Behavioral Heath Center, Charlotte, North Carolina
  - NorthCoast Clinical Trials, Inc, Beachwood, Ohio
  - Neuro-Behavioral Clinical Research, Inc, Canton, Ohio
  - Patient Priority Clinical Sites, LLC, Cinncinnati, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - NorthStar Medical Research, LLC, Middleburg Heights, Ohio
  - Summitt Research Network (Oregon), Portland, Oregon
  - Suburban Research Associates, Media, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - USC School of Medicine- Department of Neuropsychiatry and Behavioral Science, Columbia, South Carolina
  - Clinical Neurosciences Solutions, Inc., Memphis, Tennessee
  - Community Clinical Research, Inc., Austin, Texas
  - FutureSearch Clinical Trials, Austin, Texas
  - Radiant Research, Salt Lake City, Utah
  - Mood Disorders Clinic, Salt Lake City, Utah
  - Psychiatric Alliance of the Blue Ridge, Charlottesville, Virginia
  - NeuroScience, Inc., Herndon, Virginia
  - Dominion Clinical Research, Midlothian, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Summit Research Network (Seattle) LLC, Seattle, Washington
  - Northbrooke Research Center, Brown Deer, Wisconsin
  - Dean Foundation, Middleton, Wisconsin

REFERENCES:
- [Derived] Hobart M, Zhang P, Weiss C, Meehan SR, Eriksson H. Adjunctive Brexpiprazole and Functioning in Major Depressive Disorder: A Pooled Analysis of Six Randomized Studies Using the Sheehan Disability Scale. Int J Neuropsychopharmacol. 2019 Mar 1;22(3):173-179. doi: 10.1093/ijnp/pyy095. PMID 30508090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a Phase 2, multicenter, randomized, double-blind, placebo-controlled study of the safety and efficacy of OPC-34712 as adjunctive therapy in the treatment of participants with major depressive disorder. This study was conducted in the United States at 50 study centers.
Pre-assignment Details: The study consisted of a 28-day Screening period, an 8-Week single-blind placebo + Antidepressant therapy (ADT) prospective Phase A. A 6-week double-blind Randomization Phase (Phase B) or single-blind Phase A+ for those participants who did not meet criteria for randomization and a Follow-up of 30 (+2) days after the last dose of study medication.
Groups:
- OPC-34712 0.15 mg Fixed Dose: The participants received 0.15 mg/day OPC-34712 as an adjunctive therapy along with the physician assigned ADT from Week 9 to Week 14/ Early Termination.
- OPC-34712 0.5 ± 0.25 mg Low Dose: The participants received 0.50 mg OPC-34712, then 0.50 ± 0.25 mg/day as an adjunctive therapy along with the physician assigned ADT from Week 9 to Week 14/ Early Termination.
- OPC-34712 1.5 ± 0.5 mg High Dose: The participants received 1.5 mg OPC-34712, then 1.5 ± 0.50 mg/day as an adjunctive therapy along with the physician assigned ADT from Week 9 to Week 14/ Early Termination.
- Placebo: The participants received double-blind placebo as an adjunctive therapy along with the physician assigned ADT from Week 9 to Week 14/ Early Termination.
- Participants in Phase A: Participants entered Phase A (single-blind prospective treatment) during which participants had received single-blind placebo plus an open-label commercially available ADT for 8 weeks at maximally tolerated doses.
- Participants in Phase A+: Based on the response at Week 8 (in Phase A), participants were either randomized to Phase B or continued single-blind treatment in Phase A+. Participants who met the criteria for a response at Week 8 were not to be randomized into Phase B but continued to receive single-blind placebo plus the maximum tolerated dose of ADT from Week 8 for an additional 6 weeks in Phase A+.
Period: Phase A
Arm/Group | OPC-34712 0.15 mg Fixed Dose | OPC-34712 0.5 ± 0.25 mg Low Dose | OPC-34712 1.5 ± 0.5 mg High Dose | Placebo | Participants in Phase A | Participants in Phase A+
Started | 0 | 0 | 0 | 0 | 849 (850 participants entered Phase A; 849 participants were treated.) | 0
Completed | 0 | 0 | 0 | 0 | 664 | 0
Not Completed | 0 | 0 | 0 | 0 | 185 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 33 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 46 | 0
Not completed — Met withdrawal criteria | 0 | 0 | 0 | 0 | 4 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 13 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 33 | 0
Not completed — Protocol deviation | 0 | 0 | 0 | 0 | 56 | 0
Period: Phase B
Arm/Group | OPC-34712 0.15 mg Fixed Dose | OPC-34712 0.5 ± 0.25 mg Low Dose | OPC-34712 1.5 ± 0.5 mg High Dose | Placebo | Participants in Phase A | Participants in Phase A+
Started | 62 (Randomized participants.) | 120 (Randomized participants.) | 121 (Randomized participants.) | 126 (Randomized participants.) | 0 | 0
Completed | 51 | 102 | 100 | 110 | 0 | 0
Not Completed | 11 | 18 | 21 | 16 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 3 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 3 | 1 | 0 | 0
Not completed — Met Withdrawal Criteria | 3 | 3 | 6 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 3 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 3 | 3 | 0 | 0
Not completed — Protocol Deviation | 4 | 8 | 2 | 6 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 1 | 4 | 0 | 0
Period: Phase A+
Arm/Group | OPC-34712 0.15 mg Fixed Dose | OPC-34712 0.5 ± 0.25 mg Low Dose | OPC-34712 1.5 ± 0.5 mg High Dose | Placebo | Participants in Phase A | Participants in Phase A+
Started | 0 | 0 | 0 | 0 | 0 | 235
Completed | 0 | 0 | 0 | 0 | 0 | 207
Not Completed | 0 | 0 | 0 | 0 | 0 | 28
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 9
Not completed — Met withdrawal criteria | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Protocol deviation | 0 | 0 | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OPC-34712 0.15 mg Fixed Dose | OPC-34712 0.5 ± 0.25 mg Low Dose | OPC-34712 1.5 ± 0.5 mg High Dose | Placebo | Total
Number analyzed (Participants) | 62 | 120 | 121 | 126 | 429
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.9 (10.8) | 44.0 (11.8) | 43.7 (11.6) | 43.3 (11.5) | 43.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 86 | 80 | 82 | 289
  Male | 21 | 34 | 41 | 44 | 140

OUTCOME MEASURES:

1. Primary Outcome: Change From the End of Phase A (Week 8 Visit) to the End of Phase B (Week 14 Visit) in Montgomery Asberg Depression Rating Scale (MADRS) Total Score.
Description: The MADRS is utilized as the primary efficacy assessment of a participant's level of depression. The MADRS consists of 10 items, all rated on a 0 to 6 scale with 0 being the "best" rating and 6 being the "worst" rating. The MADRS Total Score is the sum of ratings for all 10 items. The possible Total scores are from 0 to 60. The MADRS Total Score was unevaluable if less than 8 of the 10 items are recorded. If 8 or 9 of the 10 items were recorded, the MADRS Total Score was the mean of the recorded items multiplied by 10 and then rounded to the first decimal place.
Time Frame: Week 8 to Week 14
Population: Intent-to-Treat (ITT) dataset consisted of all randomized participants who had an End of Phase A value and at least one post-randomization efficacy evaluation for MADRS Total Score in Phase B. The Last Observation Carried Forward (LOCF) method was used to impute missing data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | OPC-34712 0.15 mg Fixed Dose | OPC-34712 0.5 ± 0.25 mg Low Dose | OPC-34712 1.5 ± 0.5 mg High Dose | Placebo
Number analyzed (Participants) | 62 | 119 | 118 | 126
Units on a scale | -6.62 (0.99) | -6.46 (0.73) | -8.23 (0.74) | -6.09 (0.72)
Statistical Analysis 1: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; The planned sample size of 120 participants per arm will yield 80% power to detect the treatment effects at a 2-tailed significance level of 0.025. The 0.025 significance level corresponds to the second level of Hochberg's procedure for handling the two primary efficacy comparisons; Test type: Superiority or Other; p = 0.6551, ANCOVA; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-2.87 to 1.81]
Statistical Analysis 2: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7037, ANCOVA; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-2.30 to 1.55]
Statistical Analysis 3: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0303, ANCOVA; Mean Difference (Final Values) = -2.14, 95% CI 2-sided [-4.08 to -0.21]

2. Secondary Outcome: Change From End of Phase A (Week 8 Visit) to End of Phase B (Week 14 Visit) in Mean Clinical Global Impression - Severity of Illness Scale (CGI-S) Score.
Description: CGI-S items are: 0 = not assessed, 1 = normal, not at all ill, 2 = borderline mentally ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill patients. The score 0 (= not assessed) was set to missing. The CGI-S was therefore a 7-point scale from 1 through 7. CGI-S was assessed at screening, baseline and each subsequent visit from Week 1 through Week 14.
Time Frame: Week 8 to Week 14
Population: ITT dataset consisted of all randomized participants who had an End of Phase A value and at least one post-randomization efficacy evaluation for MADRS Total Score in Phase B. The LOCF method was used to impute missing data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | OPC-34712 0.15 mg Fixed Dose | OPC-34712 0.5 ± 0.25 mg Low Dose | OPC-34712 1.5 ± 0.5 mg High Dose | Placebo
Number analyzed (Participants) | 62 | 119 | 118 | 126
Units on a scale | -0.83 (0.13) | -0.81 (0.10) | -1.06 (0.10) | -0.71 (0.09)
Statistical Analysis 1: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Test type: Superiority or Other; p = 0.4166, ANCOVA; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.43 to 0.18] — Treatment difference = difference in adjusted mean change: OPC-34712 - placebo
Statistical Analysis 2: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Test type: Superiority or Other; p = 0.4193, ANCOVA; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.35 to 0.15] — Treatment difference = difference in adjusted mean change: OPC-34712 - placebo
Statistical Analysis 3: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Test type: Superiority or Other; p = 0.0064, ANCOVA; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.60 to -0.10] — Treatment difference = difference in adjusted mean change: OPC-34712 - placebo

3. Secondary Outcome: Change From End of Phase A (Week 8 Visit) to End of Phase B (Week 14 Visit) in Mean Quality of Life, Enjoyment, and Satisfaction Questionnaire - Short Form (QLES-Q-SF) Subscale Score - the Overall General Subscore (Sum of First 14 Items).
Description: The Q-LES-Q is a self-report measure to enable physicians to obtain sensitive measures of the degree of enjoyment and satisfaction experienced by participants in various areas of daily functioning. Each item is scored on a five-point scale, with 1= Very Poor; 2=Poor; 3=Fair; 4=Good; 5=Very Good. Lower scores indicating less enjoyment or satisfaction with the activity. The Overall-General Subscore will be defined by summing the scores on all 14 items and expressing it as the percent of the maximum possible score. When expressing the total score as a percentage, if items are left blank the range will be modified to reflect the number of items scored. Raw score is sum of non-missing ratings from items 1 to 14. Minimum score is number of non-missing items. Maximum score is 5*(minimum score). Range is maximum score minus minimum score. Total score is 100*(Raw score minus minimum score)/ Range, rounded to nearest integer.
Time Frame: Week 8 to Week 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of maximum possible score
Arm/Group | OPC-34712 0.15 mg Fixed Dose | OPC-34712 0.5 ± 0.25 mg Low Dose | OPC-34712 1.5 ± 0.5 mg High Dose | Placebo
Number analyzed (Participants) | 61 | 112 | 113 | 120
Percentage of maximum possible score | 7.60 (1.82) | 6.53 (1.38) | 7.46 (1.38) | 5.92 (1.34)
Statistical Analysis 1: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Test type: Superiority or Other; p = 0.4490, ANCOVA; Mean Difference (Final Values) = 1.68, 95% CI 2-sided [-2.67 to 6.02] — Treatment difference = difference in adjusted mean change: OPC-34712 - placebo
Statistical Analysis 2: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Test type: Superiority or Other; p = 0.7412, ANCOVA; Mean Difference (Final Values) = 0.61, 95% CI 2-sided [-3.02 to 4.24] — Treatment difference = difference in adjusted mean change: OPC-34712 - placebo
Statistical Analysis 3: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Test type: Superiority or Other; p = 0.4070, ANCOVA; Mean Difference (Final Values) = 1.54, 95% CI 2-sided [-2.10 to 5.17] — Treatment difference = difference in adjusted mean change: OPC-34712 - placebo

4. Secondary Outcome: Change From End of Phase A (Week 8 Visit) to End of Phase B (Week 14 Visit) in Sheehan Disability Scale (SDS) Mean Score (the Mean of 3 Individual Item Scores).
Description: The Sheehan Disability Scale (SDS) is a self-rated instrument used to measure the effect of the participant's symptoms on work/school, social life, and family/home responsibilities. For each of the three items, scores range from 0 through 10. The number most representative of how much each area was disrupted by symptoms is marked along the line from 0 = not at all, to 10 = extremely. For the work/school item, no response was to be entered if the participant did not work or go to school for reasons unrelated to the disorder and a response therefore not being applicable. The Mean SDS Score will be calculated over the three item scores. All three item scores need to be available with the exception of the work/school item score when this item is not applicable.
Time Frame: Week 8 to Week 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | OPC-34712 0.15 mg Fixed Dose | OPC-34712 0.5 ± 0.25 mg Low Dose | OPC-34712 1.5 ± 0.5 mg High Dose | Placebo
Number analyzed (Participants) | 61 | 111 | 113 | 120
Units on a scale | -0.84 (0.27) | -0.80 (0.21) | -1.27 (0.20) | -0.61 (0.20)
Statistical Analysis 1: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Test type: Superiority or Other; p = 0.4954, ANCOVA; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.86 to 0.42] — Treatment difference = difference in adjusted mean change: OPC-34712 - placebo
Statistical Analysis 2: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Test type: Superiority or Other; p = 0.4902, ANCOVA; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.73 to 0.35] — Treatment difference = difference in adjusted mean change: OPC-34712 - placebo
Statistical Analysis 3: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Test type: Superiority or Other; p = 0.0161, ANCOVA; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-1.20 to -0.12] — Treatment difference = difference in adjusted mean change: OPC-34712 - placebo

5. Secondary Outcome: Change From End of Phase A (Week 8 Visit) in MADRS Total Score for Every Study Week Visit in Phase B Other Than the Week 14 Visit.
Description: The MADRS is utilized as the primary efficacy assessment of a patient's level of depression. The MADRS consists of 10 items, all rated on a 0 to 6 scale with 0 being the "best" rating and 6 being the "worst" rating. The MADRS Total Score is the sum of ratings for all 10 items. The possible Total scores are from 0 to 60. The MADRS Total Score was unevaluable if less than 8 of the 10 items are recorded. If 8 or 9 of the 10 items were recorded, the MADRS Total Score was the mean of the recorded items multiplied by 10 and then rounded to the first decimal place.
Time Frame: Week 8 to each of Week 9, 10, 11, 12 and 13.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OPC-34712 0.15 mg Fixed Dose | OPC-34712 0.5 ± 0.25 mg Low Dose | OPC-34712 1.5 ± 0.5 mg High Dose | Placebo
Number analyzed (Participants) | 62 | 119 | 118 | 126
Units on a scale
  Week 9 (N=61,117,116,121) | -2.13 (5.22) | -3.00 (5.13) | -2.75 (5.32) | -2.48 (5.43)
  Week 10 (N=62,119,118,126) | -3.69 (5.34) | -3.78 (6.27) | -4.97 (6.48) | -3.64 (6.65)
  Week 11 (N=62,119,118,126) | -5.53 (7.24) | -5.71 (7.15) | -5.88 (7.09) | -4.40 (7.05)
  Week 12 (N=62,119,118,126) | -6.97 (7.65) | -6.31 (6.72) | -7.01 (7.58) | -4.41 (6.74)
  Week 13 (N=62,119,118,126) | -6.90 (7.71) | -6.76 (7.20) | -7.18 (7.64) | -5.47 (7.47)

6. Secondary Outcome: Change From End of Phase A (Week 8 Visit) in Mean CGI-S Score for Every Study Week Visit in Phase B Other Than the Week 14 Visit.
Description: as for outcome 2
Time Frame: Week 8 to each of Week 9, 10, 11, 12 and 13.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OPC-34712 0.15 mg Fixed Dose | OPC-34712 0.5 ± 0.25 mg Low Dose | OPC-34712 1.5 ± 0.5 mg High Dose | Placebo
Number analyzed (Participants) | 62 | 119 | 118 | 126
Units on a scale
  Week 9 (N=62,117,116,121) | -0.21 (0.60) | -0.26 (0.57) | -0.33 (0.64) | -0.21 (0.58)
  Week 10 (N=62,119,118,126) | -0.42 (0.74) | -0.39 (0.77) | -0.61 (0.91) | -0.40 (0.87)
  Week 11 (N=62,119,118,126) | -0.53 (0.95) | -0.53 (0.84) | -0.69 (0.92) | -0.47 (0.89)
  Week 12 (N=62,119,118,126) | -0.76 (1.02) | -0.66 (0.87) | -0.86 (1.00) | -0.52 (0.98)
  Week 13 (N=62,119,118,126) | -0.74 (1.09) | -0.78 (0.95) | -0.88 (1.01) | -0.59 (1.04)

7. Secondary Outcome: Change From End of Phase A (Week 8 Visit) to End of Phase B (Week 14 Visit) in Mean Q-LES-Q-SF Item 15 Score (Satisfaction With Medication).
Description: The Q-LES-Q (Short Form) is a self-report measure designed to enable physicians to easily obtain sensitive measures of the degree of enjoyment and satisfaction experienced by participants in various areas of daily functioning. Each item is scored on a five-point scale, with 1= Very Poor; 2=Poor; 3=Fair; 4=Good; 5=Very Good. Lower scores indicating less enjoyment or satisfaction with the activity. According to the scoring system suggested for this questionnaire, item 15 (Satisfaction with Medication) will yield a separate subscore.
Time Frame: Week 8 to Week 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OPC-34712 0.15 mg Fixed Dose | OPC-34712 0.5 ± 0.25 mg Low Dose | OPC-34712 1.5 ± 0.5 mg High Dose | Placebo
Number analyzed (Participants) | 61 | 111 | 113 | 120
Units on a scale | 0.02 (0.22) | 0.01 (0.25) | 0.02 (0.33) | 0.00 (0.22)

8. Secondary Outcome: Change From End of Phase A (Week 8 Visit) to End of Phase B (Week 14 Visit) in Mean Q-LES-Q-SF Item 16 Score (Overall Life Satisfaction).
Description: The Q-LES-Q (Short Form) is a self-report measure designed to enable physicians to easily obtain sensitive measures of the degree of enjoyment and satisfaction experienced by participants in various areas of daily functioning. Each item is scored on a five-point scale, with 1= Very Poor; 2=Poor; 3=Fair; 4=Good; 5=Very Good. Lower scores indicating less enjoyment or satisfaction with the activity. According to the scoring system suggested for this questionnaire, item 16 (Overall Life Satisfaction) will yield a separate subscore.
Time Frame: Week 8 to Week 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OPC-34712 0.15 mg Fixed Dose | OPC-34712 0.5 ± 0.25 mg Low Dose | OPC-34712 1.5 ± 0.5 mg High Dose | Placebo
Number analyzed (Participants) | 61 | 112 | 113 | 120
Units on a scale | 0.30 (0.84) | 0.30 (0.79) | 0.35 (0.93) | 0.28 (1.00)

9. Secondary Outcome: Change From End of Phase A (Week 8 Visit) for Every Study Week Visit in Phase B in Inventory of Depressive Symptomatology (Self-Report) (IDS-SR) Total Score.
Description: The IDS-SR is a 30-item self-report measure used to assess core diagnostic depressive symptoms as well as atypical and melancholic symptom features of major depressive disorders. The IDS-SR consists of 30 items, all rated on a 0 to 3 scale with 0 being the "best" rating and 3 being the "worst" rating. The IDS-SR Total Score is the sum of ratings of 28 item scores. The possible IDS-SR Total Score ranges from 0 to 84. The IDS-SR Total Score was un-evaluable if less than 23 of the 28 items are recorded. If the number of items was at least 23 and at most 27, the IDS-SR Total Score will be the mean of the recorded items multiplied by 28 and then rounded to the first decimal place.
Time Frame: Week 8 to each of Week 9, 10, 11, 12, 13 and 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OPC-34712 0.15 mg Fixed Dose | OPC-34712 0.5 ± 0.25 mg Low Dose | OPC-34712 1.5 ± 0.5 mg High Dose | Placebo
Number analyzed (Participants) | 62 | 119 | 118 | 126
Units on a scale
  Week 9 (N=61, 117,116,121) | -0.98 (7.28) | -1.88 (6.60) | -2.04 (5.93) | -0.98 (7.58)
  Week 10 (N=62, 119, 118, 126) | -2.13 (8.02) | -2.58 (7.37) | -4.08 (7.25) | -1.62 (7.76)
  Week 11 (N=62, 119, 118, 126) | -3.58 (7.81) | -3.41 (7.88) | -4.82 (7.96) | -2.09 (8.42)
  Week 12 (N=62, 119, 118, 126) | -5.11 (9.42) | -3.77 (8.45) | -5.77 (9.26) | -2.07 (8.42)
  Week 13 (N=62, 119, 118, 126) | -5.34 (9.15) | -5.22 (8.72) | -5.65 (8.84) | -2.37 (8.45)
  Week 14 (N=62, 119, 118, 126) | -5.55 (9.65) | -4.96 (9.37) | -6.74 (9.76) | -3.08 (9.32)

10. Secondary Outcome: Change From End of Phase A (Week 8 Visit) to End of Phase B (Week 14 Visit) in Hamilton Depression Rating Scale (HAM-D17) Score.
Description: The HAM-D17 is utilized as a secondary assessment of a participant's level of depression. The HAM-D (17-Item) consists of 17 items. Eight items are rated on a 0 to 2 scale (items 4, 5, 6, 12, 13, 14, 16 and 17), while nine items (items 1, 2, 3, 7, 8, 9, 10, 11, and 15) are rated on a 0 to 4 scale (twice the weight of the other items). For all of these items, 0 is the "best" rating and the highest score (2 or 4) is the "worst" rating. The possible total scores are from 0 to 52.
Time Frame: Week 8 to Week 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | OPC-34712 0.15 mg Fixed Dose | OPC-34712 0.5 ± 0.25 mg Low Dose | OPC-34712 1.5 ± 0.5 mg High Dose | Placebo
Number analyzed (Participants) | 48 | 98 | 101 | 109
Units on a scale | -5.77 (0.86) | -5.28 (0.63) | -6.59 (0.62) | -5.23 (0.59)
Statistical Analysis 1: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Test type: Superiority or Other; p = 0.5953, ANCOVA; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-2.54 to 1.46] — Treatment difference = difference in adjusted mean change: OPC-34712 - placebo
Statistical Analysis 2: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Test type: Superiority or Other; p = 0.9479, ANCOVA; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-1.66 to 1.55] — Treatment difference = difference in adjusted mean change: OPC-34712 - placebo
Statistical Analysis 3: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Test type: Superiority or Other; p = 0.0919, ANCOVA; Mean Difference (Final Values) = -1.36, 95% CI 2-sided [-2.95 to 0.22] — Treatment difference = difference in adjusted mean change: OPC-34712 - placebo

11. Secondary Outcome: Clinical Global Impression-Improvement Scale (CGI-I) Score at Each Study Week Visit in Phase B.
Description: CGI-I items are: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, 7 = very much worse. The score of 0 (= not assessed) will be set to missing. The CGI-I is therefore a 7-point scale from 1 through 7. CGI-I was assessed at each visit in Phase B, and improvement is judged with respect to the participant's condition at baseline. CGI-I was also assessed at each visit in Phase B, but in that phase improvement is judged with respect to the partcipant's condition at the end of Phase A.
Time Frame: Week 8 to each of Week 9, 10, 11, 12, 13 and 14.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OPC-34712 0.15 mg Fixed Dose | OPC-34712 0.5 ± 0.25 mg Low Dose | OPC-34712 1.5 ± 0.5 mg High Dose | Placebo
Number analyzed (Participants) | 62 | 119 | 118 | 126
Units on a scale
  Week 9 (N=62, 117, 116, 121) | 3.39 (0.86) | 3.30 (0.79) | 3.20 (0.80) | 3.31 (0.79)
  Week 10 (N=62, 119, 118, 126) | 3.16 (0.94) | 3.19 (0.90) | 2.95 (0.93) | 3.11 (1.04)
  Week 11 (N=62, 119, 118, 126) | 2.94 (0.94) | 3.02 (0.98) | 2.80 (0.92) | 2.94 (1.01)
  Week 12 (N=62, 119, 118, 126) | 2.87 (1.06) | 2.90 (0.99) | 2.70 (1.03) | 2.95 (1.06)
  Week 13 (N=62, 119, 118, 126) | 2.85 (1.13) | 2.76 (1.02) | 2.64 (1.06) | 2.90 (1.14)
  Week 14 (N=62, 119, 118, 126) | 2.74 (1.16) | 2.78 (1.02) | 2.52 (1.08) | 2.83 (1.12)
Statistical Analysis 1: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 9 values presented here; Test type: Superiority or Other; p = 0.3998, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel row mean scores differ test controlling for study center
Statistical Analysis 2: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 9 values presented here; Test type: Superiority or Other; p = 0.8838, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel row mean scores differ test controlling for study center
Statistical Analysis 3: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 9 values presented here; Test type: Superiority or Other; p = 0.4012, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel row mean scores differ test controlling for study center
Statistical Analysis 4: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 10 values presented here; Test type: Superiority or Other; p = 0.6131, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel row mean scores differ test controlling for study center
Statistical Analysis 5: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 10 values presented here; Test type: Superiority or Other; p = 0.5964, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel row mean scores differ test controlling for study center
Statistical Analysis 6: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 10 values presented here; Test type: Superiority or Other; p = 0.2540, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel row mean scores differ test controlling for study center
Statistical Analysis 7: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 11 values presented here; Test type: Superiority or Other; p = 0.8524, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel row mean scores differ test controlling for study center
Statistical Analysis 8: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 11 values presented here; Test type: Superiority or Other; p = 0.6969, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel row mean scores differ test controlling for study center
Statistical Analysis 9: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 11 values presented here; Test type: Superiority or Other; p = 0.3108, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel row mean scores differ test controlling for study center
Statistical Analysis 10: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 12 values presented here; Test type: Superiority or Other; p = 0.8719, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel row mean scores differ test controlling for study center
Statistical Analysis 11: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 12 values presented here; Test type: Superiority or Other; p = 0.6105, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel row mean scores differ test controlling for study center
Statistical Analysis 12: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 12 values presented here; Test type: Superiority or Other; p = 0.0709, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel row mean scores differ test controlling for study center
Statistical Analysis 13: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 13 values presented here; Test type: Superiority or Other; p = 0.9574, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel row mean scores differ test controlling for study center
Statistical Analysis 14: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 13 values presented here; Test type: Superiority or Other; p = 0.2310, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel row mean scores differ test controlling for study center
Statistical Analysis 15: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 13 values presented here; Test type: Superiority or Other; p = 0.0672, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel row mean scores differ test controlling for study center
Statistical Analysis 16: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 14 values presented here; Test type: Superiority or Other; p = 0.8441, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel row mean scores differ test controlling for study center
Statistical Analysis 17: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 14 values presented here; Test type: Superiority or Other; p = 0.6741, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel row mean scores differ test controlling for study center
Statistical Analysis 18: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 14 values presented here; Test type: Superiority or Other; p = 0.0183, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel row mean scores differ test controlling for study center

12. Secondary Outcome: Percentage of Participants With MADRS Response From End of Phase A (Week 8 Visit).
Description: A MADRS response was defined as >/= 50% reduction in MADRS Total Score from end of Phase A (Week 8 visit).
Time Frame: Week 8 to each of Week 9, 10, 11, 12, 13 and 14.
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | OPC-34712 0.15 mg Fixed Dose | OPC-34712 0.5 ± 0.25 mg Low Dose | OPC-34712 1.5 ± 0.5 mg High Dose | Placebo
Number analyzed (Participants) | 62 | 119 | 118 | 126
Percentage of participants
  Week 9 (N=61, 117, 116, 121) | 4.92 | 6.84 | 2.59 | 8.26
  Week 10 (N=62, 119, 118, 126) | 8.06 | 8.40 | 11.0 | 9.52
  Week 11 (N=62, 119, 118, 126) | 19.4 | 15.1 | 18.6 | 13.5
  Week 12 (N=62, 119, 118, 126) | 30.6 | 15.1 | 25.4 | 11.9
  Week 13 (N=62, 119, 118, 126) | 24.2 | 22.7 | 25.4 | 18.3
  Week 14 (N=62, 119, 118, 126) | 27.4 | 20.2 | 34.7 | 19.8
Statistical Analysis 1: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 9 values presented here; Test type: Superiority or Other; p = 0.3007, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 0.49, 95% CI 2-sided [0.12 to 1.93]
Statistical Analysis 2: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 9 values presented here; Test type: Superiority or Other; p = 0.8812, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 0.94, 95% CI 2-sided [0.42 to 2.10]
Statistical Analysis 3: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 9 values presented here; Test type: Superiority or Other; p = 0.0553, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 0.32, 95% CI 2-sided [0.10 to 1.07]
Statistical Analysis 4: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 10 values presented here; Test type: Superiority or Other; p = 0.6051, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 0.78, 95% CI 2-sided [0.30 to 2.05]
Statistical Analysis 5: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 10 values presented here; Test type: Superiority or Other; p = 0.8264, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 0.92, 95% CI 2-sided [0.46 to 1.85]
Statistical Analysis 6: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 10 values presented here; Test type: Superiority or Other; p = 0.8690, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 1.06, 95% CI 2-sided [0.54 to 2.10]
Statistical Analysis 7: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 11 values presented here; Test type: Superiority or Other; p = 0.3441, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 1.35, 95% CI 2-sided [0.74 to 2.44]
Statistical Analysis 8: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 11 values presented here; Test type: Superiority or Other; p = 0.6375, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 1.14, 95% CI 2-sided [0.67 to 1.94]
Statistical Analysis 9: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 11 values presented here; Test type: Superiority or Other; p = 0.3135, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 1.31, 95% CI 2-sided [0.78 to 2.21]
Statistical Analysis 10: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 12 values presented here; Test type: Superiority or Other; p = 0.0035, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 2.35, 95% CI 2-sided [1.32 to 4.18]
Statistical Analysis 11: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 12 values presented here; Test type: Superiority or Other; p = 0.4358, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 1.27, 95% CI 2-sided [0.70 to 2.31]
Statistical Analysis 12: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 12 values presented here; Test type: Superiority or Other; p = 0.0063, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 2.02, 95% CI 2-sided [1.20 to 3.41]
Statistical Analysis 13: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 13 values presented here; Test type: Superiority or Other; p = 0.3968, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 1.27, 95% CI 2-sided [0.72 to 2.23]
Statistical Analysis 14: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 13 values presented here; Test type: Superiority or Other; p = 0.2990, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 1.27, 95% CI 2-sided [0.81 to 2.00]
Statistical Analysis 15: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 13 values presented here; Test type: Superiority or Other; p = 0.1614, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 1.39, 95% CI 2-sided [0.86 to 2.25]
Statistical Analysis 16: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 14 values presented here; Test type: Superiority or Other; p = 0.3254, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 1.29, 95% CI 2-sided [0.79 to 2.12]
Statistical Analysis 17: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 14 values presented here; Test type: Superiority or Other; p = 0.9463, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 1.02, 95% CI 2-sided [0.64 to 1.62]
Statistical Analysis 18: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 14 values presented here; Test type: Superiority or Other; p = 0.0080, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 1.74, 95% CI 2-sided [1.14 to 2.65]

13. Secondary Outcome: Percentage of Participants With MADRS Remission From End of Phase A (Week 8 Visit).
Description: A MADRS remission was defined as MADRS Total Score </= 10 and >/= 50% reduction in MADRS Total Score from end of Phase A (Week 8 visit).
Time Frame: Week 8 to each of Week 9, 10, 11, 12, 13 and 14.
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | OPC-34712 0.15 mg Fixed Dose | OPC-34712 0.5 ± 0.25 mg Low Dose | OPC-34712 1.5 ± 0.5 mg High Dose | Placebo
Number analyzed (Participants) | 62 | 119 | 118 | 126
Percentage of participants
  Week 9 (N=61, 117, 116, 121) | 3.28 | 1.71 | 1.72 | 4.13
  Week 10 (N=62, 119, 118, 126) | 8.06 | 5.04 | 10.2 | 8.73
  Week 11 (N=62, 119, 118, 126) | 12.9 | 10.1 | 14.4 | 11.1
  Week 12 (N=62, 119, 118, 126) | 21.0 | 10.1 | 19.5 | 10.3
  Week 13 (N=62, 119, 118, 126) | 19.4 | 16.8 | 15.3 | 15.1
  Week 14 (N=62, 119, 118, 126) | 22.6 | 15.1 | 23.7 | 13.5
Statistical Analysis 1: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 9 values presented here; Test type: Superiority or Other; p = 0.5791, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Remission Rate = 0.59, 95% CI 2-sided [0.09 to 3.90]
Statistical Analysis 2: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 9 values presented here; Test type: Superiority or Other; p = 0.2653, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Remission Rate = 0.43, 95% CI 2-sided [0.10 to 1.93]
Statistical Analysis 3: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 9 values presented here; Test type: Superiority or Other; p = 0.2259, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Remission Rate = 0.39, 95% CI 2-sided [0.08 to 1.87]
Statistical Analysis 4: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 10 values presented here; Test type: Superiority or Other; p = 0.6986, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Remission Rate = 0.83, 95% CI 2-sided [0.32 to 2.18]
Statistical Analysis 5: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 10 values presented here; Test type: Superiority or Other; p = 0.2339, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Remission Rate = 0.61, 95% CI 2-sided [0.28 to 1.35]
Statistical Analysis 6: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 10 values presented here; Test type: Superiority or Other; p = 0.8615, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Remission Rate = 1.07, 95% CI 2-sided [0.53 to 2.15]
Statistical Analysis 7: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 11 values presented here; Test type: Superiority or Other; p = 0.8807, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Remission Rate = 1.06, 95% CI 2-sided [0.51 to 2.20]
Statistical Analysis 8: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 11 values presented here; Test type: Superiority or Other; p = 0.9035, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Remission Rate = 0.96, 95% CI 2-sided [0.52 to 1.77]
Statistical Analysis 9: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 11 values presented here; Test type: Superiority or Other; p = 0.5898, Cochran-Mantel-Haenszel; Ratio of Remission Rate = 1.19, 95% CI 2-sided [0.64 to 2.24]
Statistical Analysis 10: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 12 values presented here; Test type: Superiority or Other; p = 0.0840, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Remission Rate = 1.82, 95% CI 2-sided [0.93 to 3.58]
Statistical Analysis 11: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 12 values presented here; Test type: Superiority or Other; p = 0.9115, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Remission Rate = 0.96, 95% CI 2-sided [0.49 to 1.88]
Statistical Analysis 12: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 12 values presented here; Test type: Superiority or Other; p = 0.0522, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Remission Rate = 1.77, 95% CI 2-sided [0.98 to 3.17]
Statistical Analysis 13: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 13 values presented here; Test type: Superiority or Other; p = 0.4997, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Remission Rate = 1.24, 95% CI 2-sided [0.65 to 2.34]
Statistical Analysis 14: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 13 values presented here; Test type: Superiority or Other; p = 0.5846, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Remission Rate = 1.16, 95% CI 2-sided [0.69 to 1.93]
Statistical Analysis 15: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 13 values presented here; Test type: Superiority or Other; p = 0.9602, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Remission Rate = 0.99, 95% CI 2-sided [0.55 to 1.76]
Statistical Analysis 16: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 14 values presented here; Test type: Superiority or Other; p = 0.1254, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Remission Rate = 1.62, 95% CI 2-sided [0.87 to 3.02]
Statistical Analysis 17: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 14 values presented here; Test type: Superiority or Other; p = 0.6670, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Remission Rate = 1.13, 95% CI 2-sided [0.65 to 1.99]
Statistical Analysis 18: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 14 values presented here; Test type: Superiority or Other; p = 0.0525, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Remission Rate = 1.70, 95% CI 2-sided [0.98 to 2.93]

14. Secondary Outcome: Percentage of Participants With CGI-I Response From End of Phase A (Week 8 Visit).
Description: CGI-I response is defined as CGI-I of 1 [very much improved] or 2 [much improved].
Time Frame: Week 9, 10, 11, 12, 13 and 14.
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | OPC-34712 0.15 mg Fixed Dose | OPC-34712 0.5 ± 0.25 mg Low Dose | OPC-34712 1.5 ± 0.5 mg High Dose | Placebo
Number analyzed (Participants) | 62 | 119 | 118 | 126
percentage of participants
  Week 9 (N=62, 117, 116, 121) | 16.1 | 11.1 | 14.7 | 14.9
  Week 10 (N=62, 119, 118, 126) | 25.8 | 17.6 | 24.6 | 27.0
  Week 11 (N=62, 119, 118, 126) | 32.3 | 29.4 | 35.6 | 29.4
  Week 12 (N=62, 119, 118, 126) | 35.5 | 33.6 | 42.4 | 31.7
  Week 13 (N=62, 119, 118, 126) | 37.1 | 37.0 | 49.2 | 33.3
  Week 14 (N=62, 119, 118, 126) | 38.7 | 37.0 | 52.5 | 41.3
Statistical Analysis 1: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 9 values presented here; Test type: Superiority or Other; p = 0.9462, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 0.98, 95% CI 2-sided [0.52 to 1.84]
Statistical Analysis 2: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 9 values presented here; Test type: Superiority or Other; p = 0.4971, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 0.80, 95% CI 2-sided [0.43 to 1.49]
Statistical Analysis 3: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 9 values presented here; Test type: Superiority or Other; p = 0.8118, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 0.93, 95% CI 2-sided [0.53 to 1.63]
Statistical Analysis 4: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 10 values presented here; Test type: Superiority or Other; p = 0.8323, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 0.95, 95% CI 2-sided [0.59 to 1.53]
Statistical Analysis 5: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 10 values presented here; Test type: Superiority or Other; p = 0.0930, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 0.68, 95% CI 2-sided [0.43 to 1.08]
Statistical Analysis 6: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 10 values presented here; Test type: Superiority or Other; p = 0.5530, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 0.88, 95% CI 2-sided [0.59 to 1.32]
Statistical Analysis 7: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 11 values presented here; Test type: Superiority or Other; p = 0.8007, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 1.06, 95% CI 2-sided [0.69 to 1.61]
Statistical Analysis 8: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 11 values presented here; Test type: Superiority or Other; p = 0.8945, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 1.03, 95% CI 2-sided [0.71 to 1.49]
Statistical Analysis 9: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 11 values presented here; Test type: Superiority or Other; p = 0.3837, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 1.17, 95% CI 2-sided [0.83 to 1.64]
Statistical Analysis 10: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 12 values presented here; Test type: Superiority or Other; p = 0.7064, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 1.09, 95% CI 2-sided [0.72 to 1.63]
Statistical Analysis 11: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 12 values presented here; Test type: Superiority or Other; p = 0.7469, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 1.06, 95% CI 2-sided [0.74 to 1.52]
Statistical Analysis 12: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 12 values presented here; Test type: Superiority or Other; p = 0.0832, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 1.34, 95% CI 2-sided [0.97 to 1.86]
Statistical Analysis 13: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 13 values presented here; Test type: Superiority or Other; p = 0.6611, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 1.09, 95% CI 2-sided [0.74 to 1.61]
Statistical Analysis 14: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 13 values presented here; Test type: Superiority or Other; p = 0.4435, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 1.13, 95% CI 2-sided [0.83 to 1.56]
Statistical Analysis 15: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 13 values presented here; Test type: Superiority or Other; p = 0.0118, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 1.47, 95% CI 2-sided [1.09 to 1.98]
Statistical Analysis 16: Comparison: OPC-34712 0.15 mg Fixed Dose vs Placebo; Week 14 values presented here; Test type: Superiority or Other; p = 0.5111, Chi-squared, Corrected — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 0.89, 95% CI 2-sided [0.63 to 1.26]
Statistical Analysis 17: Comparison: OPC-34712 0.5 ± 0.25 mg Low Dose vs Placebo; Week 14 values presented here; Test type: Superiority or Other; p = 0.4903, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 0.90, 95% CI 2-sided [0.66 to 1.22]
Statistical Analysis 18: Comparison: OPC-34712 1.5 ± 0.5 mg High Dose vs Placebo; Week 14 values presented here; Test type: Superiority or Other; p = 0.0662, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel general association test controlling for study center; Ratio of Response Rate = 1.28, 95% CI 2-sided [0.98 to 1.67]

ADVERSE EVENTS:
Time Frame: From Randomization to 30 (+2) days after the end of Phase B (Week 14/End of treatment).
Description: The Safety Sample comprises those randomized participants in Phase B who received at least one dose of double-blind study medication as indicated on the dosing record.
Groups:
- OPC-34712 0.15 mg Fixed Dose: The participants received 0.15 mg/day OPC-34712 along with the physician assigned ADT from Week 9 to Week 14/ Early Termination.
- OPC-34712 0.5 ± 0.25 mg Low Dose: The participants received 0.50 mg OPC-34712, then 0.50 ± 0.25 mg/day along with the physician assigned ADT from Week 9 to Week 14/ Early Termination.
- OPC-34712 1.5 ± 0.5 mg High Dose: The participants received 1.5 mg OPC-34712, then 1.5 ± 0.50 mg/day along with the physician assigned ADT from Week 9 to Week 14/ Early Termination.
Arm/Group | OPC-34712 0.15 mg Fixed Dose | OPC-34712 0.5 ± 0.25 mg Low Dose | OPC-34712 1.5 ± 0.5 mg High Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/120 | 2/121 | 1/126
Other Adverse Events (participants affected / at risk) | 21/62 | 37/120 | 47/121 | 37/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-34712 0.15 mg Fixed Dose (N=62) | OPC-34712 0.5 ± 0.25 mg Low Dose (N=120) | OPC-34712 1.5 ± 0.5 mg High Dose (N=121) | Placebo (N=126)
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Renal mass (Renal and urinary disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-34712 0.15 mg Fixed Dose (N=62) | OPC-34712 0.5 ± 0.25 mg Low Dose (N=120) | OPC-34712 1.5 ± 0.5 mg High Dose (N=121) | Placebo (N=126)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 10 | 5
Nausea (Gastrointestinal disorders) | 0 | 7 | 2 | 3
Nasopharyngitis (Infections and infestations) | 3 | 7 | 5 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 10 | 7 | 6
Weight increased (Investigations) | 3 | 7 | 9 | 1
Akathisia (Nervous system disorders) | 4 | 6 | 10 | 4
Insomnia (Psychiatric disorders) | 5 | 3 | 4 | 4
Restlessness (Psychiatric disorders) | 4 | 1 | 5 | 6
Headache (Nervous system disorders) | 5 | 9 | 6 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No